CLINICAL TRIAL: NCT00074906
Title: Venticute in Patients With Pneumonia or Aspiration of Gastric Contents Leading to Intubation, Ventilation, and Severe Oxygenation Impairment: A Randomized, Multinational, Multicenter, Parallel Group, Double Blind, Control Group Study
Brief Title: Venticute in Patients With Pneumonia or Aspiration of Gastric Contents and Intubation/Ventilation/Oxygenation Impairment (BY2001/M1-007)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BY2001/M1-007
Record Dates: First submitted 2003-12-23; First posted 2003-12-25 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-01

CONDITIONS: Pneumonia
Keywords: Aspiration of gastric contents
MeSH Terms: conditions — Pneumonia | interventions — Venticute

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Venticute — Patients With Pneumonia or Aspiration of Gastric Contents and Intubation/Ventilation/Oxygenation Impairment

SUMMARY:
Study to demonstrate that administration of Venticute increases survival of patients with pneumonia or aspiration of gastric contents leading to intubation, mechanical ventilation, and severe oxygenation impairment.

ELIGIBILITY:
Main inclusion criteria:

* Patient has been intubated due to one of the following primary pulmonary insults: aspiration of gastric contents or pneumonia

Main exclusion criteria:

* Principal source of infection or sepsis is outside the lung
* Severe pre-existing lung disease
* Cancer metastatic to the lung or any end stage malignancy
* History of lung, liver, pancreas, small bowel, or bone marrow/stem cell transplantation
* Patient is morbidly obese
* Patient has a diagnosis of acute necrotizing pancreatitis

Additional criteria may apply and examination by an investigator is required to determine eligibility.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2003-11; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Survival on day 28 | 28 days

SECONDARY OUTCOMES:
How long the lung and the patient (overall) are recovering | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Roger G. Spragg, MD, Principal Investigator — University of California and La Jolla Veterans Affairs Medical Center, San Diego, CA, USA; Werner Seeger, MD, Principal Investigator — Justus-Liebig-Universität, Gießen, Germany; Andreas Günther, MD, Principal Investigator — University of Giessen
Locations (80):
- Australia (11):
  - Altana Pharma/Nycomed, Adelaide SA
  - Altana Pharma/Nycomed, Bedford Park, Adelaide S
  - Altana Pharma/Nycomed, Clayton, VIC
  - Altana Pharma/Nycomed, Fremantle, WA
  - Altana Pharma/Nycomed, Heidelberg, Victoria
  - Altana Pharma/Nycomed, Kingswood, Sydney, NS
  - Altana Pharma/Nycomed, Melbourne VIC
  - Altana Pharma/Nycomed, Perth, Western Australi
  - Altana Pharma/Nycomed, Southport Gold Coast QL
  - Altana Pharma/Nycomed, Victoria
  - Altana Pharma/Nycomed, Woolloongabba, Queens
- Austria (2):
  - Altana Pharma/Nycomed, Linz
  - Altana Pharma/Nycomed, Vienna
- Belgium (3):
  - Altana Pharma/Nycomed, Brussels
  - Altana Pharma/Nycomed, Edegern
  - Altana Pharma/Nycomed, Ghent
- Denmark (3):
  - Altana Pharma/Nycomed, Copenhagen NV
  - Altana Pharma/Nycomed, Hvidovre
  - Altana Pharma/Nycomed, Kolding
- Estonia (2):
  - Altana Pharma/Nycomed, Tallinn
  - Altana Pharma/Nycomed, Tartu
- Finland (6):
  - Altana Pharma/Nycomed, Jyväskylä
  - Altana Pharma/Nycomed, Kuopio
  - Altana Pharma/Nycomed, Lappeenranta
  - Altana Pharma/Nycomed, Oulu
  - Altana Pharma/Nycomed, Tampere
  - Altana Pharma/Nycomed, Turku
- Germany (12):
  - Altana Pharma/Nycomed, Berlin
  - Altana Pharma/Nycomed, Bonn
  - Altana Pharma/Nycomed, Dresden
  - Altana Pharma/Nycomed, Giessen
  - Altana Pharma/Nycomed, Greifswald
  - Altana Pharma/Nycomed, Hanover
  - Altana Pharma/Nycomed, Hofheim
  - Altana Pharma/Nycomed, Konstanz
  - Altana Pharma/Nycomed, Lübeck
  - Altana Pharma/Nycomed, München
  - Altana Pharma/Nycomed, Regensburg
  - Altana Pharma/Nycomed, Tübingen
- Greece (4):
  - Altana Pharma/Nycomed, Athens
  - Altana Pharma/Nycomed, Dragana, Alexandroupoli
  - Altana Pharma/Nycomed, Thessaloniki
  - Altana Pharma/Nycomed, Voutes, Crete
- Hungary (5):
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Kistarcsa
  - Altana Pharma/Nycomed, Szeged
  - Altana Pharma/Nycomed, Székesfehérvár
  - Altana Pharma/Nycomed, Vác
- Israel (3):
  - Altana Pharma/Nycomed, Afula
  - Altana Pharma/Nycomed, Tel Litwinsky
  - Altana Pharma/Nycomed, Ẕerifin
- Netherlands (4):
  - Altana Pharma/Nycomed, Breda
  - Altana Pharma/Nycomed, Heerlen
  - Altana Pharma/Nycomed, Rotterdam
  - Altana Pharma/Nycomed, Tilburg
- New Zealand (3):
  - Altana Pharma/Nycomed, Christchurch
  - Altana Pharma/Nycomed, Hastings
  - Altana Pharma/Nycomed, Wellington
- Altana Pharma/Nycomed, Moscow, Russia
- South Africa (2):
  - Altana Pharma/Nycomed, Johannesburg
  - Altana Pharma/Nycomed, Queenswood
- Spain (7):
  - Altana Pharma/Nycomed, Badajoz
  - Altana Pharma/Nycomed, Barcelona
  - Altana Pharma/Nycomed, Getafe (Madrid)
  - Altana Pharma/Nycomed, Granada
  - Altana Pharma/Nycomed, Madrid
  - Altana Pharma/Nycomed, Palma de Mallorca
  - Altana Pharma/Nycomed, Seville
- Switzerland (4):
  - Altana Pharma/Nycomed, Bern
  - Altana Pharma/Nycomed, Lugano
  - Altana Pharma/Nycomed, Winterthur
  - Altana Pharma/Nycomed, Zurich
- United Kingdom (8):
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Cardiff
  - Altana Pharma/Nycomed, Cottingham
  - Altana Pharma/Nycomed, Kings Lynn, Norfolk
  - Altana Pharma/Nycomed, Leeds
  - Altana Pharma/Nycomed, Nottingham
  - Altana Pharma/Nycomed, Reading
  - Altana Pharma/Nycomed, West Lothian

REFERENCES:
- [Derived] Spragg RG, Taut FJ, Lewis JF, Schenk P, Ruppert C, Dean N, Krell K, Karabinis A, Gunther A. Recombinant surfactant protein C-based surfactant for patients with severe direct lung injury. Am J Respir Crit Care Med. 2011 Apr 15;183(8):1055-61. doi: 10.1164/rccm.201009-1424OC. Epub 2010 Dec 10. PMID 21148720